CLINICAL TRIAL: NCT03449017
Title: The Effects of Electronic Cigarette Use on Alcohol Consumption: A Neurocognitive and Behavioral Investigation
Brief Title: Reactions to E-cigs and Alcohol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Alexandra Hershberger, PI, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1511771735; F31AA024682 (NIH)
Record Dates: First submitted 2018-02-21; First posted 2018-02-28 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Alcohol Abuse; Nicotine Dependence Tobacco Product
Keywords: nicotine; alcohol; vape; electronic cigarette
MeSH Terms: conditions — Alcoholism; Tobacco Use Disorder; Vaping | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Intervention Model Description: 2 session x 2 condition within participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- E-cig use condition (Experimental): Participants self-administer their own electronic cigarette device
  Interventions: Behavioral: E-cig use

INTERVENTIONS:
Behavioral: E-cig use — Self-administration of e-cig (10 puffs in 5 minutes) prior to lab task, self-administration of e-cig (10 puffs in 5 minutes) prior to ad lib alcohol, and ad lib e-cig use throughout ad lib alcohol paradigm.

SUMMARY:
The purpose of this study is to 1) examine cognitive acuity following e-cig use (as compared to no e-cig use), 2) examine motor coordination following beer and e-cig use (as compared to beer consumption only).

DETAILED DESCRIPTION:
Participants will be recruited via study fliers and notices in the community and via word-of-mouth. After viewing study advertisements, participants will call the lab and complete an over the phone screening questionnaire (approximately 10 minutes) with a trained research assistant (trained by PI, completed CITI training). If qualified participants will schedule two sessions (each approximately 4 hours for each session) to come to the lab and complete the study. Participants will receive an appointment reminder by e-mail approximately 48 hours prior to their scheduled study time. Two sessions will be scheduled (in counterbalanced order): One in which the participant will be exposed to e-cigarette cue and be allowed to use their e-cigarette during the alcohol taste test (e-cig cue session) and one in which they will not be exposed to e-cig cues or be allowed to use their e-cig during the alcohol taste test (no e-cig cue session). Participants will be asked to not schedule any sessions on days or the day before they have obligations (e.g. tests, work) in order to help ensure their participation in the study does not affect outside obligations. Participants will be paid $100 for study completion

After qualifying for the study in the phone screen, participants will complete two separate counterbalanced sessions: the e-cig cue session and the no e-cig cue session.

1. Participants will report to the lab where they will undergo informed consent process. Then, the researcher will ask the person to rinse their mouth with water and then will administer a breath alcohol test using a Breathalyzer, by asking the participant to breathe into the breathalyzer for approximately 10 seconds. The breathalyzer produces an immediate reading of BrAC. If > 0.00, a second rinse and reading will be conducted to avoid false positive readings. If positive on the second reading, participants will be excluded from the study, but the participant will not be able to leave the lab until their BrAC falls below 0.02. Participants will then be escorted to a private bathroom and will be asked to give a urine sample in a small cup. The research assistant will then use drug and pregnancy (women only) "dip stick" tests to determine pregnancy or drug use. Results are given within 2 minutes. If positive on either, a second test will be conducted on the same urine sample to avoid false positive readings. If positive again, Dr. Melissa Cyders, HSPP, who will be on call for the study, will be contacted. Dr. Cyders will use her expertise in clinical psychology and she and the research assistant will inform the participant of the positive test and provide the individual with any resources they would like (e.g. obstetrician referrals, physical examination appointment setting, drug use referrals). In case of two positive screens for pregnancy or for any drug other than marijuana, participants will be dismissed from the study. Informed consent and initial screening process takes approximately 15 minutes.
2. Participants will fill out the following surveys on a computer about their substance use and other psychological factors: The UPPS-P Impulsive Behavior Scale, the Alcohol Use Disorder Identification Test, the Nicotine and Other Substance Interaction Expectancies Questionnaire E-cig Revised, The Alcohol Expectancy Questionnaire, the Smoking Consequences Questionnaire, the Timeline Follow Back, the Fagerstrom test for Nicotine Dependence, Demographics, current e-cig craving, current alcohol craving, current mood assessment and Smoking Assessments. (approx 25 45 min)
3. Participants will complete either the e-cig cue session below or the no-e-cig cue session below (one in session 1 and the other in session 2):

   1. In the e-cig cue session, participants will be asked to bring their own e-cig and an e-cig refill liquid or cartridge. Researchers are telling participants that the study is examining the effect of nicotine use on cognitive acuity. Participants will then be asked to take 10 puffs from their e-cig over a five-minute period, consistent with findings on average puffs per use.Then, participants will report e-cig and alcohol craving and mood. Following this rating, all participants will then complete the visual dot probe task with eye tracking, using an Eye-Trac D6 Desktop mounted camera. Participants will face a computer, approximately 24 inches from the computer screen, and their eye movements will be calibrated to ensure accuracy of eye movement tracking. For the dot probe task, participants will first see a pair of alcohol-related pictures and matched control pictures, (approximately 7 x 5 inches as used in previous work) which will be presented for 1000ms. After picture offset, a visual probe appears where one of the pictures had previously been presented and participants will be instructed to identify the location of the probe as quickly as possible by pressing either the left or right mouse button. Following completion of the dot-probe tasks, participants will self-report alcohol and e-cig craving and mood (craving assessment 3) and rate the e-cig using the e-cig rating form. (eye-tracking task, including time to calibrate participants eye, takes approximately 30 minutes) Then, participants will be moved into an adjoining research room to complete what researchers are presenting as the motor coordination task. This room is equipped with a comfortable recliner, TV, and computer. Participants will be permitted to use their e-cig throughout the session and will sample 5 beers (two are non-alcoholic). Participants will be asked to self-report e-cig and alcohol craving and mood (craving assessment 4) and will then be asked to complete a beer taste test (15 minutes for technician to set up beer taste testing). The researcher will ask participants to continue to use their e-cig as they would like throughout the taste test portion of the study. Participants will be given 5 minutes prior to the beginning of the taste test to take 10 puffs of their e-cig. Prior to beginning the taste test, participants will be reminded that they will be dismissed from the study as scheduled and will have to stay for the entire allotted study time, regardless of the amount of beer they consume during the session. They will be given their beer-rating sheet and the researcher will leave the room. Participants will be unaware that the researcher, trained in session coding, will record the timing of e-cig puffs and sips of beer temporally, through the use of the lab's one-way mirror.

      Three beers with similar per volume alcohol content (Bud Light- 4.2% alcohol, Miller Light-4.2% alcohol, Sam Adams Light-4.1% alcohol) will be provided. In order to limit overall breath alcohol content of participants, Buckler's and O'Doul's (both 0% alcohol) will also be provided. All drinks will be measured (in mL) by a highly trained research assistant over the age of 21, and poured into separate cold glasses. Beers will be placed on a table in front of where the participant will be seated. In session 2, participants will be told researchers have selected their previously rated favorite beer from session 1, along with new beers to rate. Participants will be told to drink as much or as little of each beer as they like and rate each beer on various qualities (e.g., taste, aroma, drinkability), but to at least drink enough to rate each beer. Participants will be instructed that they have approximately 60 minutes to complete the taste test.

      After approximately 60 minutes, participants will have their BrAC measured (rinsing with water prior to measurement), will report their alcohol and e-cig craving and mood (craving assessment 5), and beers will be removed and measured (in mL). Participants will complete a field sobriety test which researchers are presenting as the motor coordination portion of the study. The participant's e-cig will be weighed at this time to calculate overall nicotine dose administered during the ad libitum session. Participants will be then be given access to snacks and movies and asked to remain in the room until the end of the session and their BrAC is at or below 0.02 and they show no detectable signs of intoxication on a field sobriety test. Preliminary data suggest that, on average, college students consume approximately half of the beer presented during ad lib drinking sessions. The maximum BrAC expected during the ad libitum session is approximately .05 (driving limit is .08 in the State of Indiana), with the maximum expected time of approximately 2.5 hours to return participants' BrAC to 0.02 or less (see Table 3); therefore, this is the time set across all participants. On average, participants reach a BrAC of zero after approximately 1-1.5 hours. Therefore, the researchers have set 1.25 hours as the time across all participants for the sobering up period; however, if participants BrAC is above .02 at the 1.25 hour mark, they will stay in the lab until they reach a BrAC of .02 or less.

      Participants will be allowed to use their e-cig ad libitum during the 60-minute session. Each participant will use as much or as little of the e-cig as they would like. Estimates of nicotine exposure to 18-24% nicotine content e-cigs results in .08mg/ml blood concentration over a one-hour period. Therefore, researchers expect the exposure to be in the range of ¼ - 1/5 of this amount, or, approximately 0.016-0.02 mg/ml blood concentration. Toxic levels are approximately 200 mg/ml.

      After this time has passed, participants will have their sobriety verified, and will complete a manipulation check, in which they will be asked what they believed to be the goals of the study, in order to assess for the believability of the beer taste test. Then, as the session is ending, the study technician will make conversation with the participant and will ask about what the participant did the day of the session and what s/he is doing the day after the session. This is to assess the effect of outside obligations on drinking behaviors. Participants who note significant obligations or guess study hypotheses will have their data excluded from analysis. Finally, participants will be compensated and then dismissed.
   2. In the no e-cig cue condition participants will sit for five minutes with a pencil in their hand (similar to an e-cig in size and weight). All participants will report e-cig and alcohol craving and mood (craving assessment 2) and complete the dot probe task and the beer taste test, as described above in the e-cig cue condition, except that no e-cig will be used throughout any portion of the study.
4. In session 2, participants will complete: breathalyzer, urine drug and pregnancy screen, and either the e-cig cue condition or no e-cig cue condition, as described above.
5. At the end of session 2, participants will be debriefed. Research Assistants will be thoroughly trained in handling any concerns participants may have following the test, and participants will be given study information, including contact information for the study sponsor, department, and university, as well as counseling services, if appropriate.

In order to diminish the possibility that subjects will leave before official release, the following steps will be taken: 1. Subject keys will be taken upon arrival to the session and returned upon dismissal; 2. Subjects who insist on leaving before these conditions are met will not be paid or rescheduled for further testing and their keys will not be returned if their BrAC is above 0.02, 3. Subjects will be kept in a private room that only exits into laboratory space and will be monitored appropriately by staff to avoid early self-dismissal; 4. Should a subject become belligerent or insist upon leaving when not safe, the PI will be notified to assist to ensure subject safety.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women, 21 years of age or older
* Regular alcohol use (reports at least one drink weekly - acceptability of average alcohol consumption will be made on a case by case basis by the PI)
* No current/prior severe alcohol or substance use disorder (endorsement of > 6 Alcohol/Drug Use history items on the phone screen)
* Current e-cigarette use (reports at least weekly use - acceptability of average e-cig use will be made on a case by case basis by the PI)
* Able to understand questionnaires/procedures in English
* Reports drinking beer (Yes/No on phone screen)

Exclusion Criteria:

* Pregnant/breast-feeding women (assessed via phone screen and urine screen)
* Unstable or significant medical disorders that may influence study outcome or participant safety as determined by Melissa Cyders (e.g., liver condition)
* Current/prior severe alcohol use disorder, current/prior severe substance use disorder (endorsement of > 6 Alcohol/Drug Use history items on the phone screen)
* Positive urine drug screen for amphetamines/meth-amphetamines, barbiturates, benzodiazapines, cocaine, opiates, or PCP [1-phenylcyclohexyl]
* Current mental health problems, such as depression, anxiety, post-traumatic stress disorder, bipolar disorder, or schizophrenia (self-reported at phone screen)
* Positive BrAC reading at the start of any study visit
* Court-mandated order to not drink alcohol
* Any condition that, in the judgment of the PI, could place the participant at risk or affect data validity

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2018-11-11 (Actual); Study Completion 2018-11-11 (Actual)

PRIMARY OUTCOMES:
Alcohol related attentional bias-Reaction time | Through 15 minute eye-tracking session
  -Subtracting average time to respond to alcohol stimuli from the average time to respond to non-alcohol stimuli -Faster reaction times to probes that replace alcohol-related versus control pictures are indicative of alcohol-related attentional biases
Alcohol related attentional bias-Initial orientation | Through 15 minute eye-tracking session
  -Percentage calculated based on the number of trials when gaze was initially directed at the alcohol-related picture and the total number of trials in which a fixation was made on either the alcohol-related or control picture
Alcohol related attentional bias-Delayed disengagement | Through 15 minute eye-tracking session
  Summing the total amount of time that fixations were directed at the regions of the screen occupied by the alcohol pictures and control pictures, respectively
Amount of beer consumed | 60 minutes ad libitum alcohol session
  mL of beer consumed
E-cigarette puffs | 60 minutes ad libitum alcohol session
  Number of times participant takes a hit (inhales and exhales vapor) from their e-cig.
Alcohol sips | 60 minute ad libitum alcohol session
  Number of times participant takes a drink of a beer

SECONDARY OUTCOMES:
Alcohol craving | Immediately prior to first e-cig prime, immediately following first e-cig prime , immediately prior to second e-cig prime, immediately following second e-cig prime, immediately following 60 minute ad lib session
  0 (not at all) to 10 (very much)
E-cig craving | Immediately prior to first e-cig prime, immediately following first e-cig prime , immediately prior to second e-cig prime, immediately following second e-cig prime, immediately following 60 minute ad lib session
  0 (not at all) to 10 (very much)
Timeline Followback combined e-cig and alcohol use | 30 days prior to study session
  Number of days that participant reports using their e-cig during a period of alcohol consumption
Amount of e-cig used | Pre and post 60 minute ad libitum alcohol session
  The weight (grams) of the e-cig prior to the ad libitum alcohol session minus the weight (grams) of the e-cig following the ad libitum alcohol session

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra R Hershberger, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana Univerisity Purdue University Indianapolis, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No